CLINICAL TRIAL: NCT06498622
Title: Adjuvant Treatment of Patients With High Risk of Recurrent Hepatocellular Carcinoma After Radical Surgery With Donafenib in Combination With Envafolimab: a Prospective, Multicentre, Single-arm Phase II Clinical Study
Brief Title: Adjuvant Treatment of Patients With High Risk of Recurrent Hepatocellular Carcinoma With Donafenib in Combination With Envafolimab
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Anhui Provincial Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023KY433
Record Dates: First submitted 2024-07-07; First posted 2024-07-12 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — donafenib; envafolimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Donafenib 100mg PO bid + Envafolimab 300mg IH D1 q3w (Experimental): Donafenib：100mg，PO，bid；Treatment cycle 6-12 months Envafolimab：300mg, IH，D1，q3w；Treatment cycle 6-12 months or 8-16 sessions Donafenib and Envafolimab will be administered until the disease recurrence, intolerable toxicity, death, withdrawal of consent or completion of 16 cycles of Envafolimab.
  Interventions: Drug: Donafenib + Envafolimab

INTERVENTIONS:
Drug: Donafenib + Envafolimab — Drug: Envafolimab Envafolimab 300mg IH D1 q3w Other Name: Immunotherapy, Anti-PD-L1 antibody
  Drug: Donafenib Donafenib 100mg PO bid Other Name: tyrosine kinase inhibitor, TKI

SUMMARY:
This is a multi-center, single arm study to evaluate the efficacy and safety of donafenib in combination with envafolimab treatment in patients with high risk of recurrent hepatocellular carcinoma after radical surgery.

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) is a malignant tumor with high morbidity and mortality. Surgical resection is the most important radical treatment. However, the recurrence rate is high especially in the patients with high risk of recurrence after curative resection. How to reduce postoperative recurrence and improve survival is currently a direction that is worth exploring.

Until now there is no standard postoperative adjuvant therapy. Various adjuvant treatment methods including immunotherapy, targeted therapy, TACE are being studied. This study is to explore the efficacy and safety of donafenib in combination with envafolimab treatment in HCC patients who are at high risk of recurrence after curative resection.

ELIGIBILITY:
Inclusion Criteria:

* 18-80 years old, male and female.
* Subjects voluntarily enrolled in this study and signed the informed consent, good compliance and co-operated with the follow-up.
* Primary hepatocellular carcinoma with postoperative histopathological diagnosis of HCC and negative margins.
* Presence of any of the following high-risk factors for recurrence: ① tumor size ≥5.0cm combined with microvascular invasion; ② number of tumors ≥3; ③ presence of portal vein cancer thrombus (vp1 or vp2 type).
* No recurrence of metastasis confirmed by imaging examination 3-7 weeks after surgery.
* ECOG score of 0-1.
* Expected survival ≥ 3 months.
* Child-Pugh score ≤ 7.
* Subjects with no previous antitumour therapy (except antiviral therapy)
* No extra-hepatic metastases or lymph node metastases.
* No significant abnormality in routine laboratory tests (blood test, liver and kidney function, coagulation function, etc.): (1) Criteria for routine blood tests need to be met (no blood and blood products transfusion within 14 days): a. Absolute neutrophil value (ANC) ≥ 1.5*10^9/L; b. Haemoglobin (HGB) ≥ 90g/L; c. Platelet count (PLT) ≥ 75*10^9/L. (2) Biochemical tests need to meet the following criteria: a. Serum albumin (ALB) ≥ 35g/L; b. Serum total bilirubin (TBIL) < 1.5*Upper Limit of Normal (ULN); c. Serum glutamic transaminase (AST), alanine aminotransferase (ALT) < 2.5*ULN; d. Serum creatinine ≤ 1.5*ULN.

Exclusion Criteria:

* Previous histologically/cytologically confirmed fibroplaque-containing hepatocellular carcinoma, sarcomatoid hepatocellular carcinoma, cholangiocarcinoma and other components.
* Histologically confirmed positive resection margin (R1 resection), presence of lymph node metastasis or extrahepatic metastasis.
* Previous or current malignancy other than hepatocellular carcinoma.
* History of hepatic encephalopathy or history of liver transplantation.
* Previous history of allergy to any component of the test drug: Envafolimab monoclonal antibody, donafini.
* Subjects with poorly controlled persistent postoperative pleural, abdominal or pericardial effusion.
* Previous antitumour therapy (except antiviral therapy).
* History of interstitial lung disease (except radiation pneumonitis not treated with hormones), non-infectious pneumonia.
* Presence of any active autoimmune disease or history of autoimmune disease in the subject (e.g., the following, but not limited to: autoimmune hepatitis, interstitial pneumonitis, uveitis, enterocolitis, hepatitis, pituitary gland inflammation, vasculitis, nephritis, hyperthyroidism, hypothyroidism subjects with vitiligo or asthma that has been in complete remission in childhood and does not require any intervention in adulthood may be enrolled subjects with asthma that requires medical intervention with bronchodilators cannot be included).
* Subjects who are on immunosuppressive, or systemic, or absorbable topical hormone therapy for immunosuppression (dose >10mg/day prednisone or other equipotent hormone) and continue to use it within 2 weeks prior to enrolment.
* A serious infection (CTCAE > grade 2) such as severe pneumonia, bacteraemia, or infectious co-morbidities requiring hospitalisation has occurred 4 weeks prior to the first use of study drug.
* Subjects who have experienced acute cardiovascular disease such as acute cerebral infarction, acute coronary syndrome, etc. within 1 month, with cardiovascular clinical symptoms or disease not well controlled.
* According to NYHA standard, grade III to IV cardiac insufficiency, or cardiac ultrasound examination suggests that the left ventricular ejection fraction (LVEF) <50%
* Uncontrollable hypertension with treated systolic blood pressure > 140 mmHg or diastolic blood pressure > 90 mmHg, hypertensive crisis or history of hypertensive encephalopathy
* Patients with a definite tendency to gastrointestinal bleeding, including the following: patients with locally active ulcerative lesions and fecal occult blood {(++) may not be enrolled} those with a history of black stools and vomiting of blood within 2 months.
* Those with abnormal coagulation function (INR>1.5 APTT>1.5 ULN) and bleeding tendency.
* Prolonged unhealed wounds or fractures major surgical procedures or severe traumatic injuries, fractures or ulcers within 4 weeks.
* Subjects with congenital or acquired immune deficiency (e.g., HIV-infected individuals), or active hepatitis (Hepatitis B reference: HBV DNA test value exceeds the upper limit of normal Hepatitis C reference: HCV viral titre or RNA test value exceeds the upper limit of normal).
* Patients with a history of psychotropic substance abuse that cannot be stopped or patients with mental disorders.
* Patients with concomitant illnesses that, in the investigator's judgement, are a serious hazard to patient safety or interfere with the patient's ability to complete the study.
* Pregnant women, lactating women, and women of childbearing age who are not using adequate contraception.
* In the judgement of the investigator, Patients who are not suitable for inclusion.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-07-20 (Estimated); Primary Completion 2027-05-20 (Estimated); Study Completion 2027-05-20 (Estimated)

PRIMARY OUTCOMES:
RFS | Observation period 24 months
  Recurrence Free Survival [Time Frame: Observation period 24 month] RFS was defined as the time from randomization to the first documented occurrence of local, regional, or metastatic HCC or death from any cause, whichever first occurred.

SECONDARY OUTCOMES:
OS | 24 months
  Overall Survival (OS）[Time Frame: 24 months] OS is defined as the time from the date of curative resection until death due to any cause.
2-year RFS rate | Observation period 24 months
  2-year Recurrence Free Survival Rate (2-year RFS rate) [Time Frame: Observation period 24 months] 2-year RFS rate is defined as the proportion of patients alive and free of recurrence at 2 years after curative resection.
2-year OS rate | 24 months
  2-year Overall Survival (OS）Rate [Time Frame: 24 months] 2-year RFS rate is defined as the proportion of patients alive at 2 years after curative resection.
AEs | 24 months
  Adverse Events (AEs) [ Time Frame: 24 months ] The grade of AEs and the number of patients with AEs are assessed based on CTCAE v5.0

CONTACTS AND LOCATIONS:
Overall Officials: Lianxin Liu, Principal Investigator — Anhui Provincial Hospital
Locations (2):
- China (2):
  - No.2 People's Hospital of Fuyang city, Fuyang, Anhui
  - Anhui province hospital, Hefei, Anhui

IPD SHARING:
Plan to Share IPD: No